CLINICAL TRIAL: NCT00690612
Title: An Open-label Extension Study of Candesartan Cilexetil in Hypertensive Pediatric Subjects Ages 1 to <11 Years: a Long Term Study
Brief Title: Study to Characterize the Long-term Clinical Experience of Atacand in Hypertensive Children Ages 1 to<11 Years (Hypertension in Pediatrics)
Acronym: HIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: James Hainer, MD, Sr. Director - Medical Research, Study Team Physician, AstraZeneca, LP
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2451C00006
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Hypertension
Keywords: pediatric; renal disease; high blood pressure
MeSH Terms: conditions — Hypertension; Kidney Diseases | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): investigator determines efficacious dose based on child's BP response.
  Interventions: Drug: candesartan cilexetil

INTERVENTIONS:
Drug: candesartan cilexetil — 0.05, 0.2, 0.4 mg/kg, oral solution, single daily dose
  Other Names: Atacand

SUMMARY:
The HIP study is designed to follow the clinical experience of young hypertensive children receiving candesartan cilexetil (Atacand) who are between the ages of 1 and less than 11 years old. The study is open label with no concurrent control group. To be eligible for HIP, children must have completed Study 328 without discontinuation due to a study drug-related AE and in the investigator's opinion, have an on-going clinical indication for an orally administered suspension of candesartan cilexetil to control blood pressure. Children will return to clinic every 3 months (more frequently at the investigator's discretion) for safety and efficacy evaluations. Safety will be monitored by serum chemistries, urinalyses, echocardiograms and by physical examinations at specified clinic visits. Blood pressure and heart rate will be measured at each clinic visit. Study drug is administered orally once a day. Investigators determine the efficacious dose ( 0.05 mg/kg; 0.2 mg/kg; 0.4 mg/kg) on a vist-by-vist basis depending on the child's BP response. It is anticipated that study dose will align closely with the effective anti-hypertensive dose determined in Study 328. If the child's hypertension is not well-controlled, dose adjustments up to a maximum of 0.4mg/kg/day and/or the addition of other antihypertensive medications are permitted, with the exception of other angiotensin receptor blockers. The HIP study offers eligible children up to two additional years of treatment with the liquid formulation of Atacand.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in Protocol 328 (without discontinuation due to a study drug related AE).
* Must sign an informed consent prior to initiating any stus dy procedures.
* Have, in the opinion of the investigator, an on-going clinical indication for oral liquid formulation of candesartan cilexetil to control hypertension
* Weight ≥ 10 kg and ≤ 40 kg.

Exclusion Criteria:

* Any situation, clinical condition (such as clinically significant declining renal function) or laboratory abnormality that, in the opinion of the investigator or sponsor, may interfere with the subject's participation in the study.
* Estimated glomerular filtration rate (GFR) <30 ml/min/1.73m2 for non-transplant patients and <40 ml/min/1.73m2 for transplant patients based on the Schwartz Formula (Schwartz et al 1987) as determined at enrollment into Study 328.
* Impaired liver function defined as either acute liver disease or chronic liver disease with persistently elevated liver enzyme values judged clinically significant by the investigator.
* Currently using any medications that, in the opinion of the investigator could negatively affect the subject when given together with candesartan cilexetil.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franz Schaefer, MD, Principal Investigator — University Children's Hospital, Heidelberg, Germany D69120
Locations (13):
- Belgium (2):
  - Research Site, Edegem, Belgium
  - Research Site, Ghent, Belgium
- Research Site, Strasbourg, France
- Germany (4):
  - Research Site, Erlangen
  - Research Site, Heidelberg
  - Research Site, Marburg
  - Research Site, Rostock
- Italy (2):
  - Research Site, Genova, GE
  - Research Site, Padua, PD
- Poland (2):
  - Research Site, Gda�sk
  - Research Site, Krakow
- Ukraine (2):
  - Research Site, Crimea
  - Research Site, Kyiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hypertensive children aged 1 to <11 years who had participated in the 1-year study (Protocol 328, D2451C00002-NCT00244621). First patient enrolled 17 Sep 2007 and last patient completed 9 Sep 2009 at Pediatric clinics in Europe.
Pre-assignment Details: Patients who had participated in the 1-year study (Protocol 328, D2451C00002-NCT00244621) and did not discontinue study due to a study drug-related adverse event (AE) and had an ongoing clinical indication for treatment with candesartan.
Groups:
- Atacand Candesartan Cilexetil: candesartan cilexetil (Atacand) approximately 0.05 mg/kg, 0.2 mg/kg, and 0.4 mg/kg doses administered in oral suspension form.
Period: Overall Study
Arm/Group | Atacand Candesartan Cilexetil
Started | 35
Completed | 32
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Atacand Candesartan Cilexetil
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: Years]
  <=11 years | 4.4 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Final Visit in Systolic Blood Pressure (SBP).
Description: Blood pressure response was defined as Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) less than the 95th percentile based on population height-adjusted charts for age and gender. Response rates were based on the proportion of patients meeting the criteria at each evaluation time point or the last available measure.
Time Frame: Every 3 months- baseline to final visit
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mm Hg)
Arm/Group | Atacand Candesartan Cilexetil
Number analyzed (Participants) | 35
Millimeters of Mercury (mm Hg) | -2.86 (11.97)

2. Primary Outcome: Mean Change From Baseline to Final Visit in Diastolic Blood Pressure (DBP).
Description: as for outcome 1
Time Frame: every 3 months - baseline to final visit
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atacand Candesartan Cilexetil
Number analyzed (Participants) | 35
mm Hg | -0.43 (12.26)

ADVERSE EVENTS:
Arm/Group | Atacand Candesartan Cilexetil
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atacand Candesartan Cilexetil (N=35)
Bronchopneumonia (Infections and infestations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Lymphoedema (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atacand Candesartan Cilexetil (N=35)
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 3
VOMITING (Gastrointestinal disorders) | 3
PYREXIA (General disorders) | 9
FATIGUE (General disorders) | 2
PHARYNGITIS (Infections and infestations) | 6
RHINITIS (Infections and infestations) | 6
NASOPHARYNGITIS (Infections and infestations) | 4
BRONCHITIS (Infections and infestations) | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3
VARICELLA (Infections and infestations) | 3
ACUTE TONSILLITIS (Infections and infestations) | 2
GASTROENTERITIS (Infections and infestations) | 2
INFLUENZA (Infections and infestations) | 2
OTITIS MEDIA (Infections and infestations) | 2
OTITIS MEDIA ACUTE (Infections and infestations) | 2
TONSILLITIS (Infections and infestations) | 2
URINARY TRACT INFECTION (Infections and infestations) | 2
ENURESIS (Renal and urinary disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 5
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days